CLINICAL TRIAL: NCT01048840
Title: The Natural History of Children With Gastroesophageal Reflux Disease (Ages 15 Months to 11 Years)
Brief Title: Natural History of Gastroesophageal Reflux (GER) in Children < 12 Years of Age
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Principal Investigator, Harland S. Winter, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: TAP-PediGERD; 2007-P-000907
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Subject with History of GERD: Children and adolescents ages 12-17 years, inclusive, seen at Children's Hospital, Boston or Massachusetts General Hospital between 1977 and 1990 for symptoms of GERD and also had biopsies and / or a pH probe that was positive for GERD.
- Controls with out GERD: Individuals that do not have a history of GERD or other GI problems prior to age 21 and whose date of birth are with in a year of a subjects

SUMMARY:
The goal of this project is to determine the long-term health outcome of children diagnosed with gastroesophageal reflux (GER). We are inviting subjects that were previously followed in the Pediatric GI programs at Massachusetts General and Children's Hospital, Boston. We have compiled a database of more than 200 subjects that completed diagnostic testing for GER in the 1970's and 1980's. Subjects are being contacted initially by mail using a previously approved recruitment letter. Subjects that fail to respond to this recruitment letter are called by phone. In each case, contact information has been abstracted from the Children's Hospital database. Subjects are then given the opportunity to complete a questionnaire either by phone or in hard copy. Subjects receive no compensation for their participation in this study. Subjects will be compared to controls. Controls will complete the same questionnaire as the subjects. Inclusion of potential controls will be determined by a lack of medical history of gastroenterological diseases before the age of 21 and whether the potential control was born within a year of a subject in the study. Controls will receive $25 to participate in the study.

ELIGIBILITY:
Inclusion Criteria for Subjects:

* Patients who were evaluated for GERD at the age of 12-17 years, inclusive at Children's Hospital, Boston or Massachusetts General Hospital
* Positive for GERD per biopsies or pH probe results

Inclusion Criteria for Controls:

* No GI diseases prior to age 21 including, but not limited to reflux, inflammatory bowel disease,Hirschsprung's disease
* Date of birth is within 1 year of a subject's date of birth

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The subjects will be selected from a database of patients seen at Children's Hospital, Boston or Massachusetts General Hospital between 1977 and 1990 who had biopsies or pH probe for symptoms of GERD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2004-09; Primary Completion 2010-06 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harland S Winter, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States